CLINICAL TRIAL: NCT01751555
Title: A Single-Arm Study Evaluating the Efficay and Safety of Tenofovir DF,Lamivudine and Efavirenz in Adults With HIV/HBV Coinfection
Brief Title: Efficacy and Safety of TDF+3TC+EFV in Adults With HIV/HBV Coinfection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: co-us-104-0405
Record Dates: First submitted 2012-12-14; First posted 2012-12-18 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2010-12

CONDITIONS: Hiv
Keywords: HBV co-infection ART TDF
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TDF/3TC/EFV Treatment HIV/HBV Co-infection (Experimental): TDF+3TC+EFV treatment regimen in Adults with HIV/HBV Coinfection
  Interventions: Drug: Regimen:TDF+3TC+EFV

INTERVENTIONS:
Drug: Regimen:TDF+3TC+EFV — TDF+3TC+EFV for HIV/HBV co-infection

SUMMARY:
This is a Phase 4 single-arm, post-marketing clinical trial evaluating the efficacy and safety of tenofovir disoproxil fumarate, lamivudine and efavirenz in adults with human immunodeficiency virus-1 and hepatitis B virus coinfection.

DETAILED DESCRIPTION:
HIV/HBV co-infections are frequently observed due to shared routes of transmission. TDF and 3TC are nucleotide analogues that can inhibit both HIV and HBV DNA polymerases. There is higher risk to cause drug resistance in treating HBV or HIV infection with 3TC or TDF monotherapy than combination trerapy. Combination tharapy could decreases drug resistance. China's HIV epidemic remains one of low prevalence overall, but with pockets of high infection among specific sub-populations and in some localities. China has a very high endemicity for hepatitis B too. A substantial proportion of HIV-infected individuals are co-infected with HBV. TDF + 3TC + EFV will be a common regimen for HIV/HBV co-infected Chinese individuals.

The purpose of this study of this study is to determine whether TDF will be safe for patients with HIV and HBV co-infection and the combination of TDF+3TC+EFV will suppress HIV and HBV viral load below LDL at week 48 of treatment in patients with HIV and HBV co-infeciton.This study will enroll 100 adult subjects and follow these patients for 48 weekes.There will be one enrollment visit(baseline) and visits at 2,4,8,12,24,36,48 weeks after initiation of the study regimen.

ELIGIBILITY:
Inclusion Criteria:

* Serologically-confirmed HIV and HBV infection
* Willingness to participate in a clinical trial
* No previous or current use of antiretroviral regimen
* Clinical conditions stable
* Blood creatinine less than 3 times the upper limit of normal values. HBV DNA>1000copies/ml, Tbil<34umol/L,ALT<400U/L
* With clinical indications for HAART

Exclusion Criteria:

* Patient refuses to sign the consent to participate
* Unwillingness to adhere to visit schedule or maintain adherence with medications
* Illnesses so serve as to likely require hospitalization
* With other conditions that not suitable to be enrolled will be subject to medical review

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with HIV RNA below LDL and HBV DNA below 2.3log10 copies/ml at week 48 | one year
  HIV and HBV viral load decreases in patients taking the regimen

SECONDARY OUTCOMES:
Incidence of targeted adverse events over 48 weeks | week 12,24,48
  Clinical and laboratory safety(liver, renal, hematologic)of TDF+3TC+EFV for HIV/HBV co-infected patients

OTHER OUTCOMES:
CD4+ cell count increase at week 48 | one year
  CD4+ cell count increases in patients receving the regimen

CONTACTS AND LOCATIONS:
Overall Officials: Fujie ZHANG, MD, Principal Investigator — National Center for AIDS/STD Control and Prevention, China CDC
Locations (1):
- National Center for AIDS/STD Control and Prevention, China CDC, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] G Matthews, A Avihingsanon, S Lewin, and others. Tenofovir-based Highly Active Antiretroviral Therapy (HAART) is associated with high rates of HBV DNA suppression and HBeAg seroconversion in Thai HIV-HBV coinfected patients. 59th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD 2008). San Francisco. October 31-November 4, 2008. Abstract 907. O Lada, A Gervais, M Branger, and others. De Novo Combination Therapy of Tenofovir Disoproxil Fumarate (TDF) Plus Lamivudine (LAM) or TDF Plus Emtricitabine (FTC) Is Associated With Early Virologic Response in HIV/HBV Co-Infected Patients. 59th Annual Meeting of the American Association for the Study of Liver Diseases (AASLD 2008). San Francisco. October 31-November 4, 2008. Abstract 922.
- [Derived] Wu YS, Zhang WW, Ling XM, Yang L, Huang SB, Wang XC, Wu H, Cai WP, Wang M, Wang H, Liu YF, He HL, Wei FL, Wu ZY, Zhang FJ. Efficacy and Safety of Tenofovir and Lamivudine in Combination with Efavirenz in Patients Co-infected with Human Immunodeficiency Virus and Hepatitis B Virus in China. Chin Med J (Engl). 2016 Feb 5;129(3):304-8. doi: 10.4103/0366-6999.174509. PMID 26831232